CLINICAL TRIAL: NCT03837340
Title: Large-scale Implementation of Community-based Mental Health Care for People With Severe and Enduring Mental Ill Health in Europe
Brief Title: Community-based Mental Health Care for People With Severe and Enduring Mental Ill Health
Acronym: RECOVER-E
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Special Psychiatric Hospital Kotor (Other)
Collaborators: Stichting Trimbos-Instituut (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 779362; 779362RECOVER-E H2020 (Other Grant/Funding Number: EU); U1111-1226-8617 (Other: WHO); SPH-3463/1 (Other: SPHKotor); PHI-01-8396 (Other: PHI Montenegro)
Record Dates: First submitted 2019-02-04; First posted 2019-02-12 (Actual); Last update posted 2020-03-20 (Actual); Status verified 2020-03

CONDITIONS: Severe Mental Disorders; Schizophrenia; Bipolar Disorder; Severe Depression
Keywords: Community mental health teams
MeSH Terms: conditions — Mental Disorders; Schizophrenia; Bipolar Disorder; Depression

STUDY DESIGN:
Intervention Model Description: There are two study arms- groups - both consisting of patients with SMI (severe mental illness). One group will be receiving care as usual, which in the actual setting means mostly medical treatment, without home care and assertive treatment through community based outreach teams. Another, intervention group, will be receiving assertive treatment care, with mobile assertive teams, consisting of at least three team members.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FACT (Experimental): Patients with SMI, receiving evidence-based interventions by the community mental health teams (CMHTs), inspired by the Flexible Assertive Community Treatment (FACT) service delivery model.
  Interventions: Other: CMHT
- CAU (Care as usual) (Active Comparator): Patients with SMI receiving usual care, meaning mostly medical treatment
  Interventions: Other: CAU

INTERVENTIONS:
Other: CMHT — Community mental health teams (CMHTs) delivering evidence-based interventions to people with SMI, inspired by the Flexible Assertive Community Treatment (FACT) service delivery model.
  Arms: FACT
Other: CAU — Care as usual (CAU) usually consisting of inpatient psychiatric care or outpatient care prescribing medication.
  Arms: CAU (Care as usual)

SUMMARY:
A single-blinded hybrid effectiveness-implementation trial (Type II), that both evaluates the intervention outcomes (clinical and service use outcomes) through patient-randomization in the implementation sites, as well as evaluates the implementation strategy chosen for the intervention and its impact on implementation outcomes (e.g. adoption, fidelity, acceptability and maintenance (continued implementation) of the intervention).

DETAILED DESCRIPTION:
The overall goal of the study is to contribute to improving the level of functioning and quality of life and mental health outcomes for people with severe and enduring mental ill health (SMI) (schizophrenia, bipolar disorder, depression) by adapting and upscaling the implementation of a community-based service delivery model in Montenegro.

Effectiveness component of the trial: Multidisciplinary community mental health teams for people with SMI.

The intervention condition offers flexible, assertive community treatment (FACT) in the community for people with SMI. FACT can intensify (e.g. provide more intensive treatment in the form of daily home visits, crisis care at home, more intensive evidence-based psycho-social and pharmacological treatments) or provide less intensive treatment depending on client need. It can also provide less intensive care during non-crisis periods, offering routine home treatment where a combination of psychological and pharmacological treatments (e.g. cognitive behavioral therapy, motivational interviewing, family-based interventions) are offered, as well as care processes (reviewing recovery and crisis/treatment plans, and the clients' Wellness Recovery Action Plan), and social care interventions (assistance in obtaining or maintaining employment, looking for reasonable accommodation options).

Care offered in this project in the intervention condition will be provided by a multidisciplinary community mental health team (CMHT), consisting of a diverse set of professionals including psychiatrists, psychologists, nurses, and social workers, that deliver integrated medical and social care that are focused on (symptomatic-, functional- and personal-) recovery.

CMHTs will provide home-based treatment inclusive of crisis resolution services and procedures for early recognition of sub-clinical psychosis and bipolar disorder, ACT, and intensive case management. Integrated care (i.e. health and social care interventions) will be provided to all clients. Furthermore, health and social care evidence-based interventions for severe mental illnesses will be employed during home treatment, such as family-based interventions, motivational interviewing, and cognitive behavioral therapies, combined with medication management and identifying employment (paid and unpaid options) and support in finding and maintaining this employment, (Wellness Recovery Action Plan (WRAP) recovery groups and housing opportunities.

Comparison condition: Usual care Health care settings and their providers randomized to the control condition receive usual care.

ELIGIBILITY:
Inclusion Criteria:

* Adults (ages 18-65), current service users, with severe and enduring mental ill-health, which, for clinical purposes, typically relates to diagnostic categories of bipolar disorder, severe depression, or schizophrenia. We use the following definition for SMI:

  * Presence of a psychiatric disorder that requires care and treatment (so, they are NOT in symptom remission)
  * Has severe limitations in social and community functioning (i.e. they are not in functional remission)
  * These problems are not transient (e.g. temporary, one-off) in nature (They are systematic and long-term)
  * Coordinated care provided by care networks or teams is needed to implement the treatment plan

Exclusion Criteria:

* Exclusion criteria at the patient level includes patients who do not consent to their data being collected who are part of the intervention or control conditions, those who are under the age of 18 at the start of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-01-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Changes in daily functioning | Baseline, 12 months and 18 months
  World Health Organisation Disability Assessment Schedule 2 (WHO-DAS2) measures health and disability-level of functioning in 6 domains:1.Cognition - understanding and communicating; 2.Mobility - moving and getting around; 3.Self-care - attending to one's hygiene,dressing, eating and staying alone; 4.Getting along - interacting with others; 5. Life activities - domestic responsibilities, leisure, work and school; 6.Participation in community activities,in society.The instrument is self-reporting; can be administered by a health worker if needed.Answers are distributed into 5 categories:"none","mild","moderate","severe"and"extreme or cannot do". It ends with 3 items where answers are presented as number of days (when difficulties were present). Score on any dimension ranges 0 to 7, results are depicted in a diagram which reflects relation between dimensions(the higher the score, the lower level of difficulties/better functioning) and changes over time.

SECONDARY OUTCOMES:
Change in health-related quality of life | Baseline, 12 months and 18 months
  Euro Quality of Life Index (Euro QoL 5-D 3-L). The instrument measures five dimensions:Dimension 1: Mobility; Dimension 2: Self-care;Dimension 3:Daily activities; Dimension 4: pain/discomfort; Dimension 5: Anxiety/ Depression.
  Each dimension can be rated at three levels: from no problems to major problems. The five dimensions can be summed into a descriptive health state with 11111 representing no problems in any of the five health dimensions and 33333 indicating major problems in any of the five health dimensions. Second part of the instrument is the Visual Analogue Scale to assess health status at baseline, where 0 signifies worst imaginable health state, and 100 signifies best imaginable health state.

CONTACTS AND LOCATIONS:
Overall Officials: Aleksandar Tomcuk, Principal Investigator — Special Psychiatric Hospital Kotor
Locations (1):
- ZU Specijalna bolnica za psihijatriju Dobrota Kotor, Kotor, Montenegro

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data will be shared with the coordinating institute and Heidelberg University Hospital, the two institutions that will be in charge of analyzing data from all participating project sites.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: During the project - and for a period of five years after the end of the project - each beneficiary will disseminate its results by disclosing them to the public by appropriate means as soon as possible, including scientific publications in any medium.
Access Criteria: In order to protect participant privacy, data will only be released if the request abides by national and European patient data laws and guidelines, by guidelines for use of mental health data, and by the guidelines set by each research site's ethical review board. Those requesting access to the data will be asked to verify their identity, provide information on how the data will be used, and provide information about their institutions. All requests and releases of data will be logged by the Data Protection Officer.All identifiable data will be kept confidential and will not be released.
  Data access will be limited to a need only basis. All research partners involved in RECOVER-E will have access to open data sets. As well, datasets will be made available to the European Commission or Global Alliance for Chronic Diseases on request. All de-identified data sets will be stored at the coordinating institute on password-protected, non-networked servers with limited access.

REFERENCES:
- [Derived] Shields-Zeeman L, Smit F, Wijnen B, Roth C, Wensing M, Petrea I; RECOVER-E consortium; Bolinski F, Bajraktarov S, Dedovic J, Keet R, Rojnic Kuzman M, Nakov V, Nica R, Novotni A, Tomcuk A, Djurisic T, Morales G, Rotaru Anghelescu T; RECOVER-E study. Community versus institutionalised care for people with severe mental illness in five countries in Southeast Europe: pooled analysis of five randomised trials. BMJ Glob Health. 2025 Oct 23;10(10):e018594. doi: 10.1136/bmjgh-2024-018594. PMID 41130742
- [Derived] Roth C, Wensing M, Kuzman MR, Bjedov S, Medved S, Istvanovic A, Grbic DS, Simetin IP, Tomcuk A, Dedovic J, Djurisic T, Nica RI, Rotaru T, Novotni A, Bajraktarov S, Milutinovic M, Nakov V, Zarkov Z, Dinolova R, Walters BH, Shields-Zeeman L, Petrea I. Experiences of healthcare staff providing community-based mental healthcare as a multidisciplinary community mental health team in Central and Eastern Europe findings from the RECOVER-E project: an observational intervention study. BMC Psychiatry. 2021 Oct 24;21(1):525. doi: 10.1186/s12888-021-03542-2. PMID 34689733
- [Derived] Wijnen BFM, Smit F, Uhernik AI, Istvanovic A, Dedovic J, Dinolova R, Nica R, Velickovski R, Wensing M, Petrea I, Shields-Zeeman L. Sustainability of Community-Based Specialized Mental Health Services in Five European Countries: Protocol for Five Randomized Controlled Trial-Based Health-Economic Evaluations Embedded in the RECOVER-E Program. JMIR Res Protoc. 2020 Jun 1;9(6):e17454. doi: 10.2196/17454. PMID 32476658